CLINICAL TRIAL: NCT01228773
Title: The Efficacy of Web-based, Tailored Program(Health Navigation®) for the Management of Cancer-Related Fatigue in Cancer Survivors
Brief Title: The Efficacy of Health Navigation® for Cancer-Related Fatigue in Cancer Survivors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Samsung Medical Center (Other); Seoul National University Hospital (Other); Korea University Anam Hospital (Other)
Responsible Party: Young Ho Yun. M.D., Ph.D. /Hospice & Palliative care branch, National Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCC-YoungHo
Record Dates: First submitted 2010-04-21; First posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2009-06

CONDITIONS: Cancer-related Fatigue
Keywords: Cancer Survivors, Fatigue, web-based, tailored program
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Providing tailored web-based care program(Health Navigation®), which provides various information related to the CRF.
  Web-based fatigue care program consists of 6 strategic areas (energy conservation, nutrition, exercise, sleep disturbance, pain, and distress); three areas (pain, exercise, sleep disturbance) are based on the transtheoretical model (TTM), and others (energy conservation, distress, nutrition) are based on psycho-education method or cognitive behavioral therapy. Cancer survivors who participate in the Web-based care program (Health Navigation®) will be received tailored EMS/SMS message that notify participants of the next program's news and the last program's issue etc.
  Interventions: Behavioral: Tailored web-based care program (Health Navigation®)
- B (Other): Attention control arm: Providing usual care for CRF. Three months later, as attention control, they will be provided tailored web-based care program(Health Navigation®), which provides various information related to the CRF.
  Interventions: Behavioral: Tailored web-based care program (Health Navigation®)

INTERVENTIONS:
Behavioral: Tailored web-based care program (Health Navigation®) — When intervention group participate in the Web-based care program (Health Navigation®), they can receive various information which is related with the CRF. Web-based fatigue care program consists of 6 strategic areas (energy conservation, nutrition, exercise, sleep disturbance, pain, and distress); three areas (pain, exercise, sleep disturbance) are based on the transtheoretical model (TTM), and others (energy conservation, distress, nutrition) are based on psycho-education method or cognitive behavioral therapy. Cancer survivors who participate in the Web-based care program (Health Navigation®) will be received tailored EMS/SMS message that notify participants of the next program's news and the last program's issue.
  Other Names: Non-tailored usual care service

SUMMARY:
The objective of this study is

1. to develop a web-based, tailored program for Cancer-related fatigue in cancer survivors, which is comprehensive and evidence-based,
2. to evaluate the efficacy for cancer-related fatigue as a result of participating in the Web based, tailored program(Health Navigation®) for 12 weeks
3. to evaluate the efficacy for quality of life, fatigue-related behavior, satisfaction with the treatment as a result of participating in the Web based, tailored program(health navigation®) for 12 weeks
4. to assess the efficacy of such intervention compared with usual care in cancer survivors

DETAILED DESCRIPTION:
*** Background

Cancer-related fatigue (CRF) and its impact on patients' quality of life has been increasing subject of research. Especially, cancer survivors who are complaining of fatigue (moderate - severe) should be cared.

Multidimensional characteristics of CRF were addressed in the NCCN guideline for CRF, and NCCN guideline points out the importance of behavioral approaches in managing of CRF.

NCCN guideline in 2008 suggests that 6 strategic areas (1) Energy Conservation, 2) Pain 3) Sleep disturbance 4) Distress 5) exercise, 6) Nutrition) are important issues in caring CRF in addition to the medical treatment caring chronic disease or co morbidity.

Behavioral strategy can lead those 6 areas to be effective.

However, to our knowledge, no study has examined the comprehensive fatigue management program.

The objective of this study is to develop the Web based, tailored program(Health Navigation®) for disease-free cancer patients to cope with CRF, and then evaluate the efficacy of the Web-based program(Health Navigation®).

From evidence extracted from a literature review, contents of the program was elaborated, and tailored from the TTM model. The curriculum is currently being reviewed and validated by an expert group of palliative care physician, oncologists, nurse, psychologist and health education scientists. The module will be pretested with a small number of patients, discussed in terms of feasibility and acceptance.

*** Method

To determine the efficacy of the program(Health Navigation®), a randomized controlled trial will be conducted:

After excluding patients with other causes (anemia, thyroid diseases, liver disease, co morbidities etc), 296 patients will be recruited based on statistical assumption of alpha (0.05), beta (0.20=power 80%), effect size (0.375) and drop out rate (10%).

First, they will be stratified according to their age (<50 vs. >50) and sex (male vs. female), cancer type (type 1: stomach cancer & colon cancer, type 2: Cervix & Breast cancer & Thyroid, type 3 : Lung cancer ), cancer stage (I-III) ; and then allocated to an intervention or a wait-list control group.

When intervention group participate in the Web-based care program (Health Navigation®), they can receive various information which is related with the CRF.

And Web-based fatigue care program consists of 6 strategic areas (energy conservation, nutrition, exercise, sleep disturbance, pain, and distress); three areas (pain, exercise, sleep disturbance) are based on the transtheoretical model (TTM), and others (energy conservation, distress, nutrition) are based on psycho-education method or cognitive behavioral therapy. Cancer survivors who participate in the Web-based care program (Health Navigation®) will be received tailored EMS/SMS message that notify participants of the next program's news and the last program's issue etc.

Their assistants (family member or friend) help them change their behaviors. Wait-list (control) group could not participate in the fatigue-care program (based on the Web based care program: Health Navigation®).

They could only be treated by usual care and use internet for health information. However, they can participate in the fatigue care program (Health Navigation®) after 12 weeks.

Data will be collected before randomization, after intervention, and after a follow-up of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥20, ≤65)
* moderate to severe fatigue (fatigue VAS ≥4), which persists at least 1 week in the Average Fatigue or the the Worst Fatigue
* Stage I-III
* Within 24 months of completion of primary treatment with curative intent (Surgery, radiotherapy, chemotherapy)
* Cancer survivors who are familiar with the high-speed internet and mobile phone, or cancer survivors who can participate in the web-based program with their supporter's assistance.

Exclusion Criteria:

* patients undergoing or planning surgery, radiation therapy or chemotherapy
* Major health problem which might cause fatigue or in which exercise/nutrition intervention is contraindicated at the discretion of clinician; from PAR-Q and ACSM test, cardiovascular disease(congestive heart failure, angina), pulmonary disease(chronic obstructive pulmonary disease, restrictive pulmonary disease), uncontrolled hypertension, poorly controlled diabetes and severe musculoskeletal disease and so on
* Sign of infection (body temperature ≥ 37.2℃, WBC≥11,000)
* Thrombocytopenia (platelet count ≤ 100,000/mcl)
* Anemia (Hb ≤ 10g/dL)
* SGOT or SGPT > 40 IU/L
* Creatinine > 1.4 mg/dL
* severe psychiatric disorders (psychotic disorder, major depression and so on) or suicidal tendencies
* dyspnea
* evidence of metastasis and recurrence
* ECOG(Eastern Cooperative Oncology Group) performance status of 3-4
* Not Korean speaking
* Not understanding of the study purpose and not written informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Score of fatigue Severity | 24 weeks
  BFI and FSS

SECONDARY OUTCOMES:
Mean scores of symptom scores | 24 weeks
Scores of EORTC QLQ-C30 | 24 weeks
stage of readiness | 24 weeks
  stage of readiness(physical activity, nutrition, sleep hygiene, distress, pain control, energy conservation)

CONTACTS AND LOCATIONS:
Overall Officials: Youngho Yun, Ph.D, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Cella D, Davis K, Breitbart W, Curt G; Fatigue Coalition. Cancer-related fatigue: prevalence of proposed diagnostic criteria in a United States sample of cancer survivors. J Clin Oncol. 2001 Jul 15;19(14):3385-91. doi: 10.1200/JCO.2001.19.14.3385. PMID 11454886
- [Result] Nieboer P, Buijs C, Rodenhuis S, Seynaeve C, Beex LV, van der Wall E, Richel DJ, Nooij MA, Voest EE, Hupperets P, Mulder NH, van der Graaf WT, TenVergert EM, van Tinteren H, de Vries EG. Fatigue and relating factors in high-risk breast cancer patients treated with adjuvant standard or high-dose chemotherapy: a longitudinal study. J Clin Oncol. 2005 Nov 20;23(33):8296-304. doi: 10.1200/JCO.2005.10.167. Epub 2005 Oct 11. PMID 16219926
- [Result] Bower JE, Ganz PA, Desmond KA, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol. 2000 Feb;18(4):743-53. doi: 10.1200/JCO.2000.18.4.743. PMID 10673515
- [Result] Servaes P, Verhagen S, Bleijenberg G. Determinants of chronic fatigue in disease-free breast cancer patients: a cross-sectional study. Ann Oncol. 2002 Apr;13(4):589-98. doi: 10.1093/annonc/mdf082. PMID 12056710
- [Result] Bower JE, Ganz PA, Desmond KA, Bernaards C, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in long-term breast carcinoma survivors: a longitudinal investigation. Cancer. 2006 Feb 15;106(4):751-8. doi: 10.1002/cncr.21671. PMID 16400678
- [Result] Curt GA, Breitbart W, Cella D, Groopman JE, Horning SJ, Itri LM, Johnson DH, Miaskowski C, Scherr SL, Portenoy RK, Vogelzang NJ. Impact of cancer-related fatigue on the lives of patients: new findings from the Fatigue Coalition. Oncologist. 2000;5(5):353-60. doi: 10.1634/theoncologist.5-5-353. PMID 11040270
- [Result] Patrick DL, Ferketich SL, Frame PS, Harris JJ, Hendricks CB, Levin B, Link MP, Lustig C, McLaughlin J, Reid LD, Turrisi AT 3rd, Unutzer J, Vernon SW; National Institutes of Health State-of-the-Science Panel. National Institutes of Health State-of-the-Science Conference Statement: Symptom management in cancer: pain, depression, and fatigue, July 15-17, 2002. J Natl Cancer Inst Monogr. 2004;(32):9-16. doi: 10.1093/jncimonographs/djg014. PMID 15263035
- [Result] Groopman JE. Fatigue in cancer and HIV/AIDS. Oncology (Williston Park). 1998 Mar;12(3):335-44; discussion 345-6, 351. PMID 9534184
- [Result] Vogelzang NJ, Breitbart W, Cella D, Curt GA, Groopman JE, Horning SJ, Itri LM, Johnson DH, Scherr SL, Portenoy RK. Patient, caregiver, and oncologist perceptions of cancer-related fatigue: results of a tripart assessment survey. The Fatigue Coalition. Semin Hematol. 1997 Jul;34(3 Suppl 2):4-12. PMID 9253778
- [Result] Ryan JL, Carroll JK, Ryan EP, Mustian KM, Fiscella K, Morrow GR. Mechanisms of cancer-related fatigue. Oncologist. 2007;12 Suppl 1:22-34. doi: 10.1634/theoncologist.12-S1-22. PMID 17573453
- [Result] Courneya KS, Mackey JR, Bell GJ, Jones LW, Field CJ, Fairey AS. Randomized controlled trial of exercise training in postmenopausal breast cancer survivors: cardiopulmonary and quality of life outcomes. J Clin Oncol. 2003 May 1;21(9):1660-8. doi: 10.1200/JCO.2003.04.093. PMID 12721239
- [Result] Courneya KS, Friedenreich CM, Sela RA, Quinney HA, Rhodes RE, Handman M. The group psychotherapy and home-based physical exercise (group-hope) trial in cancer survivors: physical fitness and quality of life outcomes. Psychooncology. 2003 Jun;12(4):357-74. doi: 10.1002/pon.658. PMID 12748973
- [Result] Daley AJ, Crank H, Saxton JM, Mutrie N, Coleman R, Roalfe A. Randomized trial of exercise therapy in women treated for breast cancer. J Clin Oncol. 2007 May 1;25(13):1713-21. doi: 10.1200/JCO.2006.09.5083. PMID 17470863
- [Result] Vallance JK, Courneya KS, Plotnikoff RC, Yasui Y, Mackey JR. Randomized controlled trial of the effects of print materials and step pedometers on physical activity and quality of life in breast cancer survivors. J Clin Oncol. 2007 Jun 10;25(17):2352-9. doi: 10.1200/JCO.2006.07.9988. PMID 17557948
- [Result] Dimeo F, Schwartz S, Wesel N, Voigt A, Thiel E. Effects of an endurance and resistance exercise program on persistent cancer-related fatigue after treatment. Ann Oncol. 2008 Aug;19(8):1495-1499. doi: 10.1093/annonc/mdn068. Epub 2008 Apr 1. PMID 18381369
- [Result] Cramp F, Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006145. doi: 10.1002/14651858.CD006145.pub2. PMID 18425939
- [Result] Fawzy NW. A psychoeducational nursing intervention to enhance coping and affective state in newly diagnosed malignant melanoma patients. Cancer Nurs. 1995 Dec;18(6):427-38. PMID 8564938
- [Result] Gielissen MF, Verhagen S, Witjes F, Bleijenberg G. Effects of cognitive behavior therapy in severely fatigued disease-free cancer patients compared with patients waiting for cognitive behavior therapy: a randomized controlled trial. J Clin Oncol. 2006 Oct 20;24(30):4882-7. doi: 10.1200/JCO.2006.06.8270. PMID 17050873
- [Result] Gielissen MF, Verhagen CA, Bleijenberg G. Cognitive behaviour therapy for fatigued cancer survivors: long-term follow-up. Br J Cancer. 2007 Sep 3;97(5):612-8. doi: 10.1038/sj.bjc.6603899. Epub 2007 Jul 24. PMID 17653075
- [Result] Barsevick AM, Dudley W, Beck S, Sweeney C, Whitmer K, Nail L. A randomized clinical trial of energy conservation for patients with cancer-related fatigue. Cancer. 2004 Mar 15;100(6):1302-10. doi: 10.1002/cncr.20111. PMID 15022300
- [Result] Yates P, Aranda S, Hargraves M, Mirolo B, Clavarino A, McLachlan S, Skerman H. Randomized controlled trial of an educational intervention for managing fatigue in women receiving adjuvant chemotherapy for early-stage breast cancer. J Clin Oncol. 2005 Sep 1;23(25):6027-36. doi: 10.1200/JCO.2005.01.271. PMID 16135471
- [Result] Demark-Wahnefried W, Clipp EC, McBride C, Lobach DF, Lipkus I, Peterson B, Clutter Snyder D, Sloane R, Arbanas J, Kraus WE. Design of FRESH START: a randomized trial of exercise and diet among cancer survivors. Med Sci Sports Exerc. 2003 Mar;35(3):415-24. doi: 10.1249/01.MSS.0000053704.28156.0F. PMID 12618570
- [Result] Demark-Wahnefried W, Clipp EC, Lipkus IM, Lobach D, Snyder DC, Sloane R, Peterson B, Macri JM, Rock CL, McBride CM, Kraus WE. Main outcomes of the FRESH START trial: a sequentially tailored, diet and exercise mailed print intervention among breast and prostate cancer survivors. J Clin Oncol. 2007 Jul 1;25(19):2709-18. doi: 10.1200/JCO.2007.10.7094. PMID 17602076
- [Result] Brendryen H, Kraft P. Happy ending: a randomized controlled trial of a digital multi-media smoking cessation intervention. Addiction. 2008 Mar;103(3):478-84; discussion 485-6. doi: 10.1111/j.1360-0443.2007.02119.x. PMID 18269367
- [Result] Riper H, Kramer J, Smit F, Conijn B, Schippers G, Cuijpers P. Web-based self-help for problem drinkers: a pragmatic randomized trial. Addiction. 2008 Feb;103(2):218-27. doi: 10.1111/j.1360-0443.2007.02063.x. PMID 18199300
- [Result] Vandelanotte C, Spathonis KM, Eakin EG, Owen N. Website-delivered physical activity interventions a review of the literature. Am J Prev Med. 2007 Jul;33(1):54-64. doi: 10.1016/j.amepre.2007.02.041. PMID 17572313
- [Result] Andersson G, Bergstrom J, Hollandare F, Carlbring P, Kaldo V, Ekselius L. Internet-based self-help for depression: randomised controlled trial. Br J Psychiatry. 2005 Nov;187:456-61. doi: 10.1192/bjp.187.5.456. PMID 16260822
- [Result] Wing RR, Tate DF, Gorin AA, Raynor HA, Fava JL. A self-regulation program for maintenance of weight loss. N Engl J Med. 2006 Oct 12;355(15):1563-71. doi: 10.1056/NEJMoa061883. PMID 17035649
- [Result] Svetkey LP, Stevens VJ, Brantley PJ, Appel LJ, Hollis JF, Loria CM, Vollmer WM, Gullion CM, Funk K, Smith P, Samuel-Hodge C, Myers V, Lien LF, Laferriere D, Kennedy B, Jerome GJ, Heinith F, Harsha DW, Evans P, Erlinger TP, Dalcin AT, Coughlin J, Charleston J, Champagne CM, Bauck A, Ard JD, Aicher K; Weight Loss Maintenance Collaborative Research Group. Comparison of strategies for sustaining weight loss: the weight loss maintenance randomized controlled trial. JAMA. 2008 Mar 12;299(10):1139-48. doi: 10.1001/jama.299.10.1139. PMID 18334689
- [Result] Warmerdam L, van Straten A, Cuijpers P. Internet-based treatment for adults with depressive symptoms: the protocol of a randomized controlled trial. BMC Psychiatry. 2007 Dec 19;7:72. doi: 10.1186/1471-244X-7-72. PMID 18093331
- [Result] van Bastelaar KM, Pouwer F, Cuijpers P, Twisk JW, Snoek FJ. Web-based cognitive behavioural therapy (W-CBT) for diabetes patients with co-morbid depression: design of a randomised controlled trial. BMC Psychiatry. 2008 Feb 19;8:9. doi: 10.1186/1471-244X-8-9. PMID 18284670
- [Result] Ahlberg K, Ekman T, Gaston-Johansson F, Mock V. Assessment and management of cancer-related fatigue in adults. Lancet. 2003 Aug 23;362(9384):640-50. doi: 10.1016/S0140-6736(03)14186-4. PMID 12944066
- [Result] Braun IM, Greenberg DB, Pirl WF. Evidenced-based report on the occurrence of fatigue in long-term cancer survivors. J Natl Compr Canc Netw. 2008 Apr;6(4):347-54. doi: 10.6004/jnccn.2008.0029. PMID 18433605
- [Result] Burton AW, Fanciullo GJ, Beasley RD, Fisch MJ. Chronic pain in the cancer survivor: a new frontier. Pain Med. 2007 Mar;8(2):189-98. doi: 10.1111/j.1526-4637.2006.00220.x. PMID 17305690
- [Result] Lyne ME, Coyne PJ, Watson AC. Pain management issues for cancer survivors. Cancer Pract. 2002 May-Jun;10 Suppl 1:S27-32. doi: 10.1046/j.1523-5394.10.s.1.8.x. PMID 12027966
- [Result] Roscoe JA, Morrow GR, Hickok JT, Bushunow P, Matteson S, Rakita D, Andrews PL. Temporal interrelationships among fatigue, circadian rhythm and depression in breast cancer patients undergoing chemotherapy treatment. Support Care Cancer. 2002 May;10(4):329-36. doi: 10.1007/s00520-001-0317-0. Epub 2001 Nov 28. PMID 12029433
- [Result] Berger AM, VonEssen S, Khun BR, Piper BF, Farr L, Agrawal S, Lynch JC, Higginbotham P. Feasibilty of a sleep intervention during adjuvant breast cancer chemotherapy. Oncol Nurs Forum. 2002 Nov-Dec;29(10):1431-41. doi: 10.1188/02.ONF.1431-1441. PMID 12432414
- [Result] Savard J, Simard S, Ivers H, Morin CM. Randomized study on the efficacy of cognitive-behavioral therapy for insomnia secondary to breast cancer, part I: Sleep and psychological effects. J Clin Oncol. 2005 Sep 1;23(25):6083-96. doi: 10.1200/JCO.2005.09.548. PMID 16135475
- [Result] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Result] Yun YH, Wang XS, Lee JS, Roh JW, Lee CG, Lee WS, Lee KS, Bang SM, Mendoza TR, Cleeland CS. Validation study of the korean version of the brief fatigue inventory. J Pain Symptom Manage. 2005 Feb;29(2):165-72. doi: 10.1016/j.jpainsymman.2004.04.013. PMID 15733808
- [Result] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Result] Yun YH, Mendoza TR, Heo DS, Yoo T, Heo BY, Park HA, Shin HC, Wang XS, Cleeland CS. Development of a cancer pain assessment tool in Korea: a validation study of a Korean version of the brief pain inventory. Oncology. 2004;66(6):439-44. doi: 10.1159/000079497. PMID 15452372
- [Result] Shim EJ, Shin YW, Jeon HJ, Hahm BJ. Distress and its correlates in Korean cancer patients: pilot use of the distress thermometer and the problem list. Psychooncology. 2008 Jun;17(6):548-55. doi: 10.1002/pon.1275. PMID 17957764
- [Result] Gessler S, Low J, Daniells E, Williams R, Brough V, Tookman A, Jones L. Screening for distress in cancer patients: is the distress thermometer a valid measure in the UK and does it measure change over time? A prospective validation study. Psychooncology. 2008 Jun;17(6):538-47. doi: 10.1002/pon.1273. PMID 17973237
- [Result] Guigoz Y, Vellas B, Garry PJ. Assessing the nutritional status of the elderly: The Mini Nutritional Assessment as part of the geriatric evaluation. Nutr Rev. 1996 Jan;54(1 Pt 2):S59-65. doi: 10.1111/j.1753-4887.1996.tb03793.x. No abstract available. PMID 8919685
- [Result] Read JA, Crockett N, Volker DH, MacLennan P, Choy ST, Beale P, Clarke SJ. Nutritional assessment in cancer: comparing the Mini-Nutritional Assessment (MNA) with the scored Patient-Generated Subjective Global Assessment (PGSGA). Nutr Cancer. 2005;53(1):51-6. doi: 10.1207/s15327914nc5301_6. PMID 16351506
- [Result] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Result] Yun YH, Mendoza TR, Kang IO, You CH, Roh JW, Lee CG, Lee WS, Lee KS, Bang SM, Park SM, Cleeland CS, Wang XS. Validation study of the Korean version of the M. D. Anderson Symptom Inventory. J Pain Symptom Manage. 2006 Apr;31(4):345-52. doi: 10.1016/j.jpainsymman.2005.07.013. PMID 16632082